CLINICAL TRIAL: NCT06274047
Title: PROSTATE-IQ: Parallel RandOmized STudy of Personalized Apalutamide Treatment and Evaluation to Improve Quality of Life in Post-Operative Radiation With Androgen Axis Suppression. A Phase III Multi-center Study for Men With Detectable PSA After Prostatectomy for Prostate Cancer.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0409; NCI-2024-01553 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Androgen Axis Suppression; Prostatectomy; Prostate Cancer
Keywords: Prostate; Salvage Radiation; ADT; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Participants will receive 6 months of standard-of-care androgen deprivation therapy (ADT) and radiation therapy.
  Interventions: Drug: Androgen Deprivation Therapy
- Arm 2 (Experimental): Participants will receive 6 months of apalutamide and radiation therapy.
  Interventions: Drug: Apalutamide
- Arm 3 (Experimental): Participants will receive 24 months of standard-of-care androgen deprivation therapy (ADT) and radiation therapy.
  Interventions: Drug: Androgen Deprivation Therapy
- Arm 4 (Experimental): Participants will receive 6 months of ADT, apalutamide, and radiation therapy.
  Interventions: Drug: Apalutamide; Drug: Androgen Deprivation Therapy

INTERVENTIONS:
Drug: Apalutamide — Given by PO
  Arms: Arm 2; Arm 4
Drug: Androgen Deprivation Therapy — Given by PO
  Other Names: ADT
  Arms: Arm 1; Arm 3; Arm 4

SUMMARY:
1. Personalize treatment for prostate cancer based on how aggressive the disease is and
2. Learn if apalutamide-based treatment can help to reduce fatigue and other side effects of treatment in participants who are being treated with radiation therapy for prostate cancer, as compared to standard therapy.

DETAILED DESCRIPTION:
Primary Objective:

ARTERA LOW COHORT (less aggressive disease)

1) To compare fatigue at 9 months, as assessed by FACIT-F, between participants assigned to six months of apalutamide monotherapy versus six months of GnRH-based ADT.

HIGHER RISK COHORT (more aggressive disease)

1) To compare fatigue at 24 months, as assessed by FACIT-fatigue, between participants assigned to six months of GnRH-based ADT plus apalutamide monotherapy versus 24 months of GnRH-based ADT.

Secondary Objectives for both Cohorts:

1. To compare patient-reported quality of life for the two treatment arms (Arm 1 vs. 2 for Artera-Low Cohort and Arm 3 vs. 4 for Artera-High Cohort) as measured by FACT-P and EPIC-26.
2. To compare physician-reported toxicity for the two treatment arms as measured by CTCAE v 5.
3. To compare patient-reported activity levels for the two treatment arms as measured by the leisure-time activity questionnaire.
4. To compare patient activity and sleep for the two treatment arms as measured by participant wearable health bands.
5. To compare cognitive function for the two treatment arms as measured by PROMIS-CF and the Symbol Digit Modality test.
6. To compare mental health for the two treatment arms as measured by the Health Anxiety and Depression Scale.
7. To compare changes in HgA1c and Lipid profiles over time between the two treatment arms.
8. To compare time to testosterone recovery between treatment arms.
9. To compare time to next therapy between treatment arms.
10. To compare progression-free survival, metastasis-free survival, cancer specific mortality and overall survival between treatment arms.
11. To compare risk of major acute coronary event between treatment arms.
12. In the subset of patients who agree to optional body composition measurements, to compare change in body composition including visceral fat and skeletal muscle mass between treatment arms.

Exploratory Objectives for both Cohorts:

1. In the subset of participants who agree to correlative studies, to evaluate the association between fatigue and circulating inflammatory cytokines.
2. In the subset of participants who agree to germline testing, to determine if inherited variants in steroidogenic genes influence individual body composition toxicity with androgen signaling inhibition.
3. To evaluate how germline variants interact with tumor intrinsic properties (via Artera) to determine the overall benefit patients derive from finite, intense androgen signaling inhibition in the post-operative setting.
4. To investigate the relationship between plasma exosomes, Artera tissue pattern, and the germline to somatic interaction.
5. To study the overlap between body composition toxicity and risk for coronary artery disease as measured by radiographic coronary calcifications and lab markers of coronary artery disease.
6. To evaluate the association between radiation plan metrics and patient-reported urinary and bowel functional changes.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate cancer.
2. PSA ≥ 0.1 after radical prostatectomy.
3. Candidate for salvage radiation and ADT treatment, as determined by treating physician.
4. Age >18 at the time of consent.
5. ECOG Performance Status ≤ 2.
6. Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 90 days of registration.

   System Laboratory Value

   Hematological:

   Platelet count (plt) = ≥ 100,000/µL

   Hemoglobin (Hgb) = ≥ 9 g/dL

   Renal:

   eGFR = ≥ 30 mL/min using MDRD Formula

   Hepatic and Other:

   Bilirubin2 = ≤1.5 x upper limit of normal (ULN) Aspartate aminotransferase (AST) = ≤ 2.5 x ULN Alanine aminotransferase (ALT) = ≤ 2.5 x ULN Serum Albumin = > 3.0 g/dL Serum potassium = ≥ 3.5 mmol/L 2In subjects with Gilbert's syndrome, if total bilirubin is >1.5 x ULN, measure direct and indirect bilirubin; if direct bilirubin is ≤ 1.5 x ULN, subject may be eligible.
7. Ability to understand and comply with study procedures for the entire length of the study as determined by the site investigator or protocol designee.
8. Ability to understand English or Spanish language as determined by the site investigator or protocol designee. Since the primary outcome is a questionnaire available in English and Spanish.
9. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately. Participants must have the ability to understand and willingness to sign the written informed consent document.

Exclusion Criteria:

1. Use of post-prostatectomy testosterone suppression prior to registration (use of GnRH agonist or antagonist, with or without an anti-androgen). However, participants with testosterone recovery after post-prostatectomy testosterone suppression are eligible (testosterone recovery defined as total testosterone > 190 ng/dL) regardless of how long their testosterone was suppressed.
2. History of any of the following:

   * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year prior to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy).
   * Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization. Any condition that in the opinion of the investigator, would preclude participation in this study.
3. Current evidence of any of the following:

   * Uncontrolled hypertension (consistently >160 systolic or >100 diastolic)
   * Gastrointestinal disorder affecting absorption
   * Active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis).
   * Any condition that in the opinion of the investigator, would preclude participation in this study.
4. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
5. Confirmed extrapelvic or bone disease
6. Medications known to lower the seizure threshold (listed in section 5 below) must be discontinued or substituted 4 weeks prior to C1D1 of study treatment for participants on arms receiving apalutamide.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue) | Through study completion; an average of 1 year.
  Score scale ranges (0-4) 0 - Not at all
  1. - A little bit
  2. - Somewhat
  3. - Quite a bit
  4. - Very Much

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hoffman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org